CLINICAL TRIAL: NCT01218880
Title: Phase I Study of M2ES Combined Gemcitabine in Patients With Advanced Pancreatic Cancer
Brief Title: Study With M2ES and Gemcitabine for Patients With Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protgen Ltd (Industry)
Responsible Party: Guodong Chang, Protgen Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2ES2010-1
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- M2ES-A (Experimental)
  Interventions: Drug: M2ES 7.5mg
- M2ES-B (Experimental)
  Interventions: Drug: M2ES 15mg
- M2ES-C (Experimental)
  Interventions: Drug: M2ES 30mg
- M2ES-D (Experimental)
  Interventions: Drug: M2ES 45mg

INTERVENTIONS:
Drug: M2ES 7.5mg — M2ES Dosage：7.5mg/m2
  Other Names: M2ES
  Arms: M2ES-A
Drug: M2ES 15mg — M2ES Dosage：15mg/m2
  Other Names: M2ES
  Arms: M2ES-B
Drug: M2ES 30mg — M2ES Dosage：30mg/m2
  Other Names: M2ES
  Arms: M2ES-C
Drug: M2ES 45mg — M2ES Dosage：45mg/m2
  Other Names: M2ES
  Arms: M2ES-D

SUMMARY:
Phase I trail will be conducted to evaluate the safety of M2ES in combination with gemcitabine in locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Phase I trail will be conducted to determine the MTD and safety of M2ES(administered intravenous infusion on Days 1,8,15,21of a 28-day cycle) in combination with gemcitabine (1000 m/m2). Gemcitabine will be administered as an intravenous infusion on Days 1, 8, and 15 of each 28-day cycle,at the same time determine the safety and efficiency of this combined regime.

ELIGIBILITY:
Inclusion Criteria:

1. patients had histologically or cytologically confirmed pancreatic adenocarcinoma that was not amenable to potentially curative surgery.
2. No prior chemotherapy was allowed.
3. Prior radiation therapy was allowed provided that the only sites of measurable disease were not located within the radiation port.
4. 18 to 60 years of age
5. Karnofsky performance status (KPS) of 60-100 points
6. Unidimensionally measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
7. Adequate hematologic, renal, and hepatic function was required as deWned by the following: WBC ≥4×109/L, absolute neutrophil count ≥ 1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥ 9g/dL, total bilirubin ≤2 upper limit of normal [ULN],AST ≤ 1.5 ULN, or ≤ 3 ULN if there was evidence of liver metastases; alkaline phosphatase ≤ 1.5 ULN, or ≤ 3 ULN if there was evidence of liver Metastases; creatinine clearance ≥50 mL/min.
8. life expectancy of at least 12 weeks.
9. All patients provided written informed consent according to federal and institutional guidelines.

Exclusion Criteria:

1. patients had clinically apparent CNS disease ( primary brain tumors, tumor related apoplexy, CNS metastases, carcinomatous meningitis.)
2. another active malignancy, or any history of other malignancy within the past 5 years except for nonmelanoma skin cancer and carcinoma in situ of the cervix.
3. more than 4 weeks intervals between the last administration of the targeted therapy regimen and study entry.
4. radiation therapy have not been completed 4 weeks before enrollment.
5. major surgery within the prior 4 weeks;
6. participating any clinical trial within the prior 4 weeks;
7. Pregnant or lactating women.
8. tumor involvement of major blood vessels
9. uncontrolled intercurrent illness as following: prior or ongoing uncontrolled hypertension;angina pectoris; congestive cardiac failure; myocardial ischemia, infarction, uncompensated coronary artery disease within the past 6 months; Uncontrolled arrhythmia; Uncontrolled diabetes mellitus; Uncontrolled infection.
10. chronic renal disease.
11. urine protein ≥ 500 mg in 24 hours;
12. prior history of gastrointestinal bleeding, hemoptysis, bleeding diathesis.
13. pulmonary embolus, or deep venous thrombosis
14. ECG: QTC ≥ 480 ms
15. Patients on therapeutic doses of heparin or antiplatelet agents.
16. Patients who received thrombolytic agents or who required full-dose anticoagulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerant dose | 8 week

SECONDARY OUTCOMES:
objective response rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhaosheng Li, MD, Principal Investigator — Shanghai Changhai Hosptial
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China